CLINICAL TRIAL: NCT02874742
Title: Phase 2, Randomized, Open-Label Study Comparing Daratumumab, Lenalidomide, Bortezomib, and Dexamethasone (D-RVd) Versus Lenalidomide, Bortezomib, and Dexamethasone (RVd) in Subjects With Newly Diagnosed Multiple Myeloma Eligible for High-Dose Chemotherapy and Autologous Stem Cell Transplantation
Brief Title: Study Comparing Daratumumab, Lenalidomide, Bortezomib, and Dexamethasone (D-RVd) Versus Lenalidomide, Bortezomib, and Dexamethasone (RVd) in Subjects With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108195; 54767414MMY2004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-08-01; First posted 2016-08-22 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Daratumumab+Lenalidomide+Bortezomib+Dexamethasone (D-RVd) (Experimental): Participants will receive lenalidomide, bortezomib, dexamethasone and daratumumab.
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone; Drug: Daratumumab
- Lenalidomide+Bortezomib+Dexamethasone (RVd) (Experimental): Participants will receive lenalidomide, bortezomib and dexamethasone.
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Cycles 1 through 6: lenalidomide 25 (milligram) mg orally on Days 1 through 14 and each cycle is of 21-days followed by maintenance treatment with lenalidomide 10 mg on days 1-21 throughout each 28-day cycle on Cycles 7 through 9. Beginning at Cycle 10, the lenalidomide dose will be increased to 15 mg unless there is a tolerability concern.
Drug: Bortezomib — Bortezomib 1.3 mg/m^2 subcutaneously on Days 1, 4, 8, and 11 during Cycles 1-6.
Drug: Dexamethasone — Dexamethasone 40 mg orally every week (20 mg on Days 1, 2, 8, 9, 15, and 16).
Drug: Daratumumab — Daratumumab intravenously at a dose of 16 milligram per kilogram (mg/kg) weekly during induction treatment (Days 1, 8, and 15 of Cycles 1 through 4), and every 3 weeks during consolidation treatment (Day 1 of Cycles 5 and 6), followed by maintenance treatment with daratumumab every 4 or 8 weeks.
  Arms: Daratumumab+Lenalidomide+Bortezomib+Dexamethasone (D-RVd)

SUMMARY:
The purpose of this study is to determine if the addition of daratumumab to lenalidomide-bortezomib-dexamethasone (RVd) will increase the proportion of participants achieving stringent complete response (sCR), as defined by the International Myeloma Working Group (IMWG) criteria, by the time of completion of post autologous stem cell transplantation (ASCT) consolidation treatment, compared with RVd alone.

ELIGIBILITY:
Inclusion Criteria:

* Considered by the investigator to be eligible for high-dose chemotherapy (HDT) and autologous stem cell transplantation (ASCT) according to the institution's criteria based on age, medical history, cardiac and pulmonary status, overall health and condition, co-morbid condition(s), physical examination, and laboratory studies
* Has not had prior systemic therapy for multiple myeloma. An emergency course of steroids (defined as no greater than 40 milligram [mg] of dexamethasone, or equivalent per day for a maximum of 4 days (that is, a total of 160 mg) is permitted. In addition, radiation therapy is permitted prior to study entry, during screening, and during Cycles 1-2 of study treatment as needed for lytic bone disease
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Woman of childbearing potential must have 2 negative highly sensitive serum (beta-human chorionic gonadotropin [b-hCG]) during screening, the first one within 10 to 14 days prior to the first dose of any component of study treatment and the second within 24 hours prior to the first dose of any component of study treatment
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study (including during dose interruptions), and for 4 weeks following discontinuation of lenalidomide, and if receiving daratumumab, for 3 months after the last dose

Exclusion Criteria:

* Diagnosed or treated for malignancy other than multiple myeloma, except: a) Malignancy treated with curative intent and with no known active disease present for more than equal to (>= )3 years before randomization; b) Adequately treated non-melanoma skin cancer, lentigo maligna or in situ malignancies (including but not limited to, cervical, breast) with no evidence of disease
* Exhibiting clinical signs of or has a known history of meningeal or central nervous system involvement by multiple myeloma
* Known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) less than (<)50 percent (%) of predicted normal
* Known moderate or severe persistent asthma within the past 2 years or currently has uncontrolled asthma of any classification
* Known to be seropositive for human immunodeficiency virus, known to have hepatitis B surface antigen positivity, or known to have a history of hepatitis C. Participants who completed treatment for hepatitis C at least 6 months prior to screening and have no detectable circulating hepatitis C virus (HCV) at screening, may participate in the study. Such participants will be required to undergo regular assessment for HCV reactivation during their participation in the study. Participants who test positive for HCV at any time during these assessments will be withdrawn from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (36):
- United States (36):
  - Birmingham, Alabama
  - Duarte, California
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Westwood, Kansas
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Buffalo, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Abington, Pennsylvania
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Voorhees PM, Sborov DW, Laubach J, Kaufman JL, Reeves B, Rodriguez C, Silbermann R, Costa LJ, Anderson LD Jr, Nathwani N, Shah N, Bumma N, Efebera YA, Holstein SA, Costello C, Jakubowiak A, Wildes TM, Orlowski RZ, Shain KH, Cowan AJ, Dinner S, Gries KS, Pei H, Cortoos A, Patel S, Lin TS, Usmani SZ, Richardson PG. A plain language summary of the final analysis of the GRIFFIN study of daratumumab plus lenalidomide, bortezomib, and dexamethasone for people with newly diagnosed multiple myeloma. Future Oncol. 2025 Jan;21(1):25-49. doi: 10.1080/14796694.2024.2408909. Epub 2024 Oct 25. PMID 39452950
- [Derived] Sonneveld P, Dimopoulos MA, Boccadoro M, Quach H, Ho PJ, Beksac M, Hulin C, Antonioli E, Leleu X, Mangiacavalli S, Perrot A, Cavo M, Belotti A, Broijl A, Gay F, Mina R, van de Donk NWCJ, Katodritou E, Schjesvold F, Balari AS, Rosinol L, Delforge M, Roeloffzen W, Silzle T, Vangsted A, Einsele H, Spencer A, Hajek R, Jurczyszyn A, Lonergan S, Ahmadi T, Liu Y, Wang J, Vieyra D, van Brummelen EMJ, Vanquickelberghe V, Sitthi-Amorn A, de Boer CJ, Carson R, Rodriguez-Otero P, Blade J, Moreau P. A plain language summary of the PERSEUS study of daratumumab plus bortezomib, lenalidomide, and dexamethasone for treating newly diagnosed multiple myeloma. Future Oncol. 2024;20(38):3043-3063. doi: 10.1080/14796694.2024.2394323. Epub 2024 Sep 17. PMID 39287147
- [Derived] Chari A, Kaufman JL, Laubach J, Sborov DW, Reeves B, Rodriguez C, Silbermann R, Costa LJ, Anderson LD Jr, Nathwani N, Shah N, Bumma N, Holstein SA, Costello C, Jakubowiak A, Wildes TM, Orlowski RZ, Shain KH, Cowan AJ, Pei H, Cortoos A, Patel S, Lin TS, Voorhees PM, Usmani SZ, Richardson PG. Daratumumab in transplant-eligible patients with newly diagnosed multiple myeloma: final analysis of clinically relevant subgroups in GRIFFIN. Blood Cancer J. 2024 Jul 8;14(1):107. doi: 10.1038/s41408-024-01088-6. PMID 38977707
- [Derived] Callander NS, Silbermann R, Kaufman JL, Godby KN, Laubach J, Schmidt TM, Sborov DW, Medvedova E, Reeves B, Dhakal B, Rodriguez C, Chhabra S, Chari A, Bal S, Anderson LD Jr, Dholaria BR, Nathwani N, Hari P, Shah N, Bumma N, Holstein SA, Costello C, Jakubowiak A, Wildes TM, Orlowski RZ, Shain KH, Cowan AJ, Pei H, Cortoos A, Patel S, Lin TS, Giri S, Costa LJ, Usmani SZ, Richardson PG, Voorhees PM. Daratumumab-based quadruplet therapy for transplant-eligible newly diagnosed multiple myeloma with high cytogenetic risk. Blood Cancer J. 2024 Apr 22;14(1):69. doi: 10.1038/s41408-024-01030-w. PMID 38649340
- [Derived] Silbermann R, Laubach J, Kaufman JL, Sborov DW, Reeves B, Rodriguez C, Chari A, Costa LJ, Anderson LD Jr, Nathwani N, Shah N, Bumma N, Holstein SA, Costello C, Jakubowiak A, Orlowski RZ, Shain KH, Cowan AJ, Gries KS, Pei H, Cortoos A, Patel S, Lin TS, Voorhees PM, Usmani SZ, Richardson PG. Health-related quality of life in transplant-eligible patients with newly diagnosed multiple myeloma treated with daratumumab, lenalidomide, bortezomib, and dexamethasone: Patient-reported outcomes from GRIFFIN. Am J Hematol. 2024 Jul;99(7):1257-1268. doi: 10.1002/ajh.27326. Epub 2024 Apr 15. PMID 38622840
- [Derived] Voorhees PM, Sborov DW, Laubach J, Kaufman JL, Reeves B, Rodriguez C, Chari A, Silbermann R, Costa LJ, Anderson LD Jr, Nathwani N, Shah N, Bumma N, Efebera YA, Holstein SA, Costello C, Jakubowiak A, Wildes TM, Orlowski RZ, Shain KH, Cowan AJ, Dinner S, Pei H, Cortoos A, Patel S, Lin TS, Usmani SZ, Richardson PG. Addition of daratumumab to lenalidomide, bortezomib, and dexamethasone for transplantation-eligible patients with newly diagnosed multiple myeloma (GRIFFIN): final analysis of an open-label, randomised, phase 2 trial. Lancet Haematol. 2023 Oct;10(10):e825-e837. doi: 10.1016/S2352-3026(23)00217-X. Epub 2023 Sep 11. PMID 37708911
- [Derived] Nooka AK, Kaufman JL, Rodriguez C, Jakubowiak A, Efebera Y, Reeves B, Wildes T, Holstein SA, Anderson LD Jr, Badros A, Shune L, Chari A, Pei H, Cortoos A, Patel S, Lin TS, Richardson PG, Voorhees P. A plain language summary of daratumumab plus lenalidomide/bortezomib/dexamethasone in transplant-eligible Black patients with newly diagnosed multiple myeloma in the GRIFFIN study. Future Oncol. 2022 Dec;18(40):4443-4456. doi: 10.2217/fon-2022-0775. Epub 2023 Feb 17. PMID 36799429
- [Derived] Sborov DW, Baljevic M, Reeves B, Laubach J, Efebera YA, Rodriguez C, Costa LJ, Chari A, Silbermann R, Holstein SA, Anderson LD Jr, Kaufman JL, Shah N, Pei H, Patel S, Cortoos A, Bartlett JB, Vermeulen J, Lin TS, Voorhees PM, Richardson PG. Daratumumab plus lenalidomide, bortezomib and dexamethasone in newly diagnosed multiple myeloma: Analysis of vascular thrombotic events in the GRIFFIN study. Br J Haematol. 2022 Nov;199(3):355-365. doi: 10.1111/bjh.18432. Epub 2022 Sep 16. PMID 36111391
- [Derived] Swan D, Henderson R, McEllistrim C, Naicker SD, Quinn J, Cahill MR, Mykytiv V, Lenihan E, Mulvaney E, Nolan M, Parker I, Natoni A, Lynch K, Ryan AE, Szegezdi E, Krawczyk J, Murphy P, O'Dwyer M. CyBorD-DARA in Newly Diagnosed Transplant-Eligible Multiple Myeloma: Results from the 16-BCNI-001/CTRIAL-IE 16-02 Study Show High Rates of MRD Negativity at End of Treatment. Clin Lymphoma Myeloma Leuk. 2022 Nov;22(11):847-852. doi: 10.1016/j.clml.2022.07.011. Epub 2022 Jul 21. PMID 35985959
- [Derived] Voorhees PM, Rodriguez C, Reeves B, Nathwani N, Costa LJ, Lutska Y, Bobba P, Hoehn D, Pei H, Ukropec J, Qi M, Lin TS, Richardson PG. Daratumumab plus RVd for newly diagnosed multiple myeloma: final analysis of the safety run-in cohort of GRIFFIN. Blood Adv. 2021 Feb 23;5(4):1092-1096. doi: 10.1182/bloodadvances.2020003642. PMID 33606004
- [Derived] Voorhees PM, Kaufman JL, Laubach J, Sborov DW, Reeves B, Rodriguez C, Chari A, Silbermann R, Costa LJ, Anderson LD Jr, Nathwani N, Shah N, Efebera YA, Holstein SA, Costello C, Jakubowiak A, Wildes TM, Orlowski RZ, Shain KH, Cowan AJ, Murphy S, Lutska Y, Pei H, Ukropec J, Vermeulen J, de Boer C, Hoehn D, Lin TS, Richardson PG. Daratumumab, lenalidomide, bortezomib, and dexamethasone for transplant-eligible newly diagnosed multiple myeloma: the GRIFFIN trial. Blood. 2020 Aug 20;136(8):936-945. doi: 10.1182/blood.2020005288. PMID 32325490

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 223 participants were enrolled/randomized (16 in safety run-in,104 to D-RVd and 103 to RVd group). Among 207 (D-RVd [104]+RVd [103]) randomized, 201 received treatment (D-RVd: 100 and RVd: 101). 1 participant randomized to D-RVd group received RVd treatment and was randomized twice (resulting a total of 224 participants).
Pre-assignment Details: Participant was a screen-failure but was mistakenly randomized first to D-RVd ; after re-screening was randomized to RVd group. The participant was counted in D-RVd for ITT analysis and RVd for safety analysis. So, safety analysis set included 99 participants in D-RVd and 102 in RVd group who received at least 1 dose of study treatment.
Groups:
- Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd): Induction and Consolidation Phase (12-week induction phase followed by autologous stem cell mobilization, high-dose chemotherapy [HDT] and autologous stem cell transplantation [ASCT]; 6-week consolidation phase)- participants received lenalidomide 25 milligrams (mg) orally on Days 1 to 14 of Cycles 1 through 6), bortezomib 1.3 mg per meter square (mg/m^2) subcutaneously (SC) on Days 1, 4, 8, and 11 and dexamethasone 40 mg orally weekly (20 mg on Days 1, 2, 8, 9, 15 and 16); Maintenance phase (up to 104 week [until disease progression/up to maximum of 2 years])- participants received lenalidomide 10 mg orally on Days 1 to 21 throughout each 28-day cycle on Cycles 7 through 9 during maintenance treatment. Beginning at Cycle 10, lenalidomide dose was increased to 15 mg, unless there was tolerability concern. After 2 years of maintenance therapy, participants could continue to lenalidomide monotherapy per standard of care. Long-term follow-up phase- all participants were followed for at least 1 year after last dose of study drug and to continue until death, withdrawal of consent or end of study.
- Randomized: Daratumumab+RVd (D-RVd): Induction and Consolidation Phase (12 week induction phase followed by autologous stem cell mobilization, HDT and ASCT; a 6-week consolidation phase)-participants received RVd with daratumumab 16 milligrams per kilogram (mg/kg) intravenously (IV) weekly on Days 1, 8, and 15 of Cycles 1 to 4 during induction treatment and every 3 weeks on Day 1 of Cycles 5 and 6 during consolidation treatment; Maintenance phase (up to 104-week [until disease progression/up to maximum of 2 years])- participants received daratumumab 16 mg/kg every 4 weeks/8 weeks plus lenalidomide 10 mg orally on Days 1 to 21 throughout each 28-day cycle on Cycles 7 through 9 during maintenance treatment. Beginning at Cycle 10, the lenalidomide dose was increased to 15 mg, unless there was a tolerability concern. After 2 years of maintenance therapy, participants could continue to lenalidomide monotherapy per standard of care. Long-term follow-up phase- all participants were followed for at least 1 year after last dose of study drug and to continue until death, withdrawal of consent or end of study. Per protocol amendment 4, to provide flexibility and prioritize safety during the global coronavirus-19 (COVID-19) pandemic, participants were given the option to switch from daratumumab IV to daratumumab SC at the discretion of the investigator.
- Safety Run-in: D-RVd: Induction and Consolidation Phase (12 week induction phase followed by autologous stem cell mobilization, HDT and ASCT; a 6-week consolidation phase)-participants received RVd with daratumumab 16 mg/kg IV weekly on Days 1, 8, and 15 of Cycles 1 to 4 during induction treatment and every 3 weeks on Day 1 of Cycles 5 and 6 during consolidation treatment; Maintenance phase (up to 104-week [until disease progression/up to maximum of 2 years])- participants received daratumumab 16 mg/kg every 4 weeks/8 weeks plus lenalidomide 10 mg orally on Days 1 to 21 throughout each 28-day cycle on Cycles 7 through 9 during maintenance treatment. Beginning at Cycle 10, the lenalidomide dose was increased to 15 mg, unless there was a tolerability concern. After 2 years of maintenance therapy, participants could continue to lenalidomide monotherapy per standard of care. Long-term follow-up phase- all participants were followed for at least 1 year after last dose of study drug and to continue until death, withdrawal of consent or end of study.
Period: Overall Study
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Started | 103 | 104 | 16
Treated (Safety Analysis Set) | 101 | 100 | 16
Completed | 76 | 88 | 15
Not Completed | 27 | 16 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 5 | 4 | 1
Not completed — Withdrawal by Subject | 17 | 8 | 0
Not completed — Other | 4 | 1 | 0
Not completed — Progressive Disease | 1 | 0 | 0
Not completed — Screen Failure | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd | Total
Number analyzed (Participants) | 103 | 104 | 16 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (7.27) | 57.2 (9.79) | 59.8 (5.96) | 58.2 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 46 | 8 | 97
  Male | 60 | 58 | 8 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Black or African American | 18 | 14 | 4 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 76 | 85 | 11 | 172
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 5 | 3 | 0 | 8
  Other | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 103 | 104 | 16 | 223

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Stringent Complete Response (sCR)
Description: Percentage of participants who had achieved sCR as determined by the validated computer algorithm according to the International Myeloma Working Group (IMWG) criteria, by the end of post-autologous stem cell transplantation (post-ASCT) consolidation treatment were reported. Complete response (CR) is defined as negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas, and less than (<) 5 percent (%) PCs in bone marrow. sCR is defined as in addition to CR a normal FLC ratio, and absence of clonal plasma cells (PCs) by immunohistochemistry or immunofluorescence or 2 to 4-color flow cytometry.
Time Frame: From randomization to post-ASCT consolidation (after Cycle 6) before maintenance treatment (up to 10 months)
Population: Response-evaluable analysis set included all participants who had a confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit, received at least 1 dose of study treatment and had at least 1 post baseline disease assessment. The outcome measure was planned to be reported for randomized participants only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd)
Number analyzed (Participants) | 97 | 99
Percentage of participants | 32.0 [22.9 to 42.2] | 42.4 [32.5 to 52.8]

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Better
Description: CR or better rate is defined as the percentage of participants who achieve CR or sCR, according to the IMWG criteria. CR is negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas, and < 5% PCs in bone marrow. sCR is defined as in addition to CR a normal FLC ratio, and absence of clonal plasma cells (PCs) by immunohistochemistry or immunofluorescence or 2 to 4-color flow cytometry. For 2 participants (1 in each randomized treatment group), data were updated by the study sites which resulted in their inclusion to the response-evaluable analysis set after the primary analysis.
Time Frame: From randomization to end of following: induction treatment, ASCT, post-ASCT consolidation (after Cycle 6) and at the end of maintenance period of 24 months (overall duration up to 34 months)
Population: Response-evaluable analysis set included all participants who had a confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit, received at least 1 dose of study treatment and had at least 1 post baseline disease assessment. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 98 | 100 | 16
Percentage of participants
  At the end of induction prior to ASCT: number analyzed (Participants) | 97 | 99 | 16
  At the end of induction prior to ASCT | 13.4 [7.3 to 21.8] | 19.2 [12.0 to 28.3] | 12.5 [1.6 to 38.3]
  At the end of ASCT prior to consolidation: number analyzed (Participants) | 97 | 99 | 16
  At the end of ASCT prior to consolidation | 19.6 [12.2 to 28.9] | 27.3 [18.8 to 37.1] | 56.3 [29.9 to 80.2]
  At the end of post-ASCT consolidation: number analyzed (Participants) | 97 | 99 | 16
  At the end of post-ASCT consolidation | 42.3 [32.3 to 52.7] | 51.5 [41.3 to 61.7] | 68.8 [41.3 to 89.0]
  At the end of maintenance period (up to 24 Months) | 60.2 [49.8 to 70.0] | 83.0 [74.2 to 89.8] | 93.8 [69.8 to 99.8]

3. Secondary Outcome: Percentage of Participants With Overall Stringent Complete Response (sCR)
Description: Overall sCR rate is defined as the percentage of participants who achieved sCR, according to the IMWG criteria. CR is defined as negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas, and < 5 % PCs in bone marrow. sCR is defined as in addition to CR a normal FLC ratio, and absence of clonal PCs by immunohistochemistry or immunofluorescence or 2 to 4-color flow cytometry.
Time Frame: From randomization to end of following: induction treatment, ASCT, post-ASCT consolidation (after Cycle 6) and at the end of maintenance treatment of 24 months (overall duration up to 34 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 98 | 100 | 16
Percentage of participants
  At the end of induction prior to ASCT: number analyzed (Participants) | 97 | 99 | 16
  At the end of induction prior to ASCT | 7.2 [3.0 to 14.3] | 12.1 [6.4 to 20.2] | 0 [NA to NA] — Here NA signifies that 95% CI was not estimable as zero participant had events during at the end of induction prior to ASCT.
  At the end of ASCT prior to consolidation: number analyzed (Participants) | 97 | 99 | 16
  At the end of ASCT prior to consolidation | 14.4 [8.1 to 23.0] | 21.2 [13.6 to 30.6] | 43.8 [19.8 to 70.1]
  At the end of post-ASCT consolidation: number analyzed (Participants) | 97 | 99 | 16
  At the end of post-ASCT consolidation | 32.0 [22.9 to 42.2] | 42.4 [32.5 to 52.8] | 56.3 [29.9 to 80.2]
  At the end of Maintenance Treatment (up to 24 Months) | 48.0 [37.8 to 58.3] | 67.0 [56.9 to 76.1] | 93.8 [69.8 to 99.8]

4. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR)
Description: ORR- percentage of participants who achieved partial response (PR) or better (PR, Very Good Partial Response [VGPR], CR or sCR) based on computerized algorithm as per IMWG criteria. PR -greater than or equal to (>=) 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg//24 hours. If serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required. A >=50% reduction in the size of soft tissue plasmacytomas is also required; VGPR-serum and urine M-component detectable by immunofixation but not on electrophoresis, or >= 90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours; CR-negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow. sCR- in addition to CR a normal FLC ratio, and absence of clonal PCs by immunohistochemistry or immunofluorescence or 2 to 4-color flow cytometry.
Time Frame: as for outcome 3
Population: Response-evaluable analysis set included all participants who had a confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit, received at least 1 dose of study treatment and had at least 1 post baseline disease assessment. Here, 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 98 | 100 | 16
Percentage of participants
  At the end of induction prior to ASCT: number analyzed (Participants) | 97 | 99 | 16
  At the end of induction prior to ASCT | 91.8 [84.4 to 96.4] | 98.0 [92.9 to 99.8] | 100 [79.4 to 100]
  At the end of ASCT prior to consolidation: number analyzed (Participants) | 97 | 99 | 16
  At the end of ASCT prior to consolidation | 91.8 [84.4 to 96.4] | 99.0 [94.5 to 100] | 100 [79.4 to 100]
  At the end of post-ASCT consolidation: number analyzed (Participants) | 97 | 99 | 16
  At the end of post-ASCT consolidation | 91.8 [84.4 to 96.4] | 99.0 [94.5 to 100] | 100 [79.4 to 100]
  At the End of Maintenance Treatment (up to 24 Months) | 91.8 [84.5 to 96.4] | 99.0 [94.6 to 100.0] | 100.0 [79.4 to 100.0]

5. Secondary Outcome: Percentage of Participants Who Achieved Very Good Partial Response (VGPR) or Better
Description: VGPR or better rate is defined as the percentage of participants who achieved VGPR or better, according to the IMWG criteria. VGPR is defined as serum and urine M-component detectable by immunofixation but not on electrophoresis, or >= 90% reduction in serum M-protein plus urine M-protein <100 mg/24 hours.
Time Frame: as for outcome 2
Population: Population analyzed included response evaluable analysis set who achieved response (PR or better). Here, 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 98 | 100 | 16
Percentage of participants
  At the end of induction prior to ASCT: number analyzed (Participants) | 97 | 99 | 16
  At the end of induction prior to ASCT | 56.7 [46.3 to 66.7] | 71.7 [61.8 to 80.3] | 68.8 [41.3 to 89.0]
  At the end of ASCT prior to consolidation: number analyzed (Participants) | 97 | 99 | 16
  At the end of ASCT prior to consolidation | 66.0 [55.7 to 75.3] | 86.9 [78.6 to 92.8] | 100 [79.4 to 100]
  At the end of post-ASCT consolidation: number analyzed (Participants) | 97 | 99 | 16
  At the end of post-ASCT consolidation | 73.2 [63.2 to 81.7] | 90.9 [83.4 to 95.8] | 100 [79.4 to 100]
  At the End of Maintenance Period (up to 24 Months) | 77.6 [68.0 to 85.4] | 96.0 [90.1 to 98.9] | 100.0 [79.4 to 100.0]

6. Secondary Outcome: Percentage of Participants With Negative Minimal Residual Disease (MRD)
Description: Minimal residual disease negative rate is defined as the percentage of participants who achieve MRD negative status by the respective time point. Minimal residual disease was evaluated in participants who achieved CR or sCR (including participants with VGPR or better and suspected daratumumab interference) using next-generation sequencing which utilizes multiple myeloma cell DNA from bone marrow aspirates at a threshold of less than (<) 10^5.
Time Frame: From randomization to end of following: induction treatment, post-ASCT consolidation (after Cycle 6) (up to 4.5 months), and at the end of maintenance period of 24 months (overall duration up to 34 months)
Population: Intent to treat (ITT) analysis set which included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 103 | 104 | 16
Percentage of participants
  MRD from randomization to prior to ASCT (10^5) | 7.8 [3.4 to 14.7] | 22.1 [14.6 to 31.3] | 18.8 [4.0 to 45.6]
  Post ASCT consolidation (10^5) | 20.4 [13.1 to 29.5] | 50.0 [40.0 to 60.0] | 50.0 [24.7 to 75.3]
  At the End of Maintenance Period (up to 24 Months) (10^5) | 30.1 [21.5 to 39.9] | 64.4 [54.4 to 73.6] | 81.3 [54.4 to 96.0]

7. Secondary Outcome: Duration of Complete Response or Better
Description: Duration of CR or better is the duration from the date of initial documentation of a CR or sCR response, according to the IMWG criteria, to the date of first documented evidence of progressive disease (PR), or relapse from CR. PD is defined as an increase of 25 % from the lowest response value in one of the following: serum and urine M-component (absolute increase must be greater than or equal to [>=] 0.5 gram per deciliter [g/dL] and >=200 milligrams [mg]/24 hours respectively); Only in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels (absolute increase must be > 10 mg/dL); Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to plasma cells (PCs) proliferative disorder.
Time Frame: From randomization to the date of first documented evidence of progressive disease or relapse from CR (up to 5 years)
Population: Population analyzed included response evaluable analysis set who achieved response (PR or better).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 90 | 99 | 16
Months | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events.

8. Secondary Outcome: Duration of Stringent Complete Response (sCR)
Description: Duration of sCR is the duration from the date of initial documentation of a sCR response, according to the IMWG criteria, to the date of first documented evidence of progressive disease, or relapse from sCR. PD is defined as an increase of 25 % from the lowest response value in one of the following: serum and urine M component (absolute increase must be >= 0.5 g/dL and >=200 mg/24 hours respectively); Only in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels (absolute increase must be > 10 mg/dL); Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: From randomization to the date of first documented evidence of progressive disease or relapse from sCR (up to 5 years)
Population: Population analyzed included response evaluable analysis set who achieved response PR or better.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 90 | 99 | 16
Months | NA [NA to NA] — Here NA signifies Median and 95% CI was not estimable due to an insufficient number of events. | NA [NA to NA] — Here NA signifies Median and 95% CI was not estimable due to an insufficient number of events. | NA [42.4 to NA] — Here NA signifies Median and 95% CI was not estimable due to an insufficient number of events.

9. Secondary Outcome: Time to Stringent Complete Response (sCR)
Description: Time to sCR is the duration from the date of randomization to the date of initial documentation of sCR, which was confirmed by a repeated measurement as required by the IMWG criteria.
Time Frame: From randomization to the date of initial documentation of sCR (up to 5 years)
Population: Response-evaluable analysis set included all participants who had a confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit, received at least 1 dose of study treatment and had at least 1 post baseline disease assessment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 98 | 100 | 16
Months | 14.3 [9.2 to 21.7] | 10.2 [8.8 to 13.0] | 8.4 [7.1 to 15.2]

10. Secondary Outcome: Time to Complete Response or Better
Description: Time to CR or better is the duration from the date of randomization to the date of initial documentation of CR or better, which was confirmed by a repeated measurement as required by the IMWG criteria.
Time Frame: From randomization to the date of initial documentation of CR (up to 5 years)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 98 | 100 | 16
Months | 9.6 [8.4 to 12.2] | 8.9 [7.9 to 9.4] | 7.7 [6.7 to 9.7]

11. Secondary Outcome: Time to Very Good Partial Response (VGPR) or Better
Description: Time to VGPR or better is the duration from the date of randomization to the date of initial documentation of VGPR or better, which was confirmed by a repeated measurement as required by the IMWG criteria.
Time Frame: From randomization to the date of initial documentation of VGPR or better (up to 5 years)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 98 | 100 | 16
Months | 3.0 [2.2 to 6.3] | 2.2 [2.1 to 2.7] | 2.1 [0.9 to 6.7]

12. Secondary Outcome: Time to Partial Response (PR) or Better
Description: Time to PR or better is the duration from the date of randomization to the date of initial documentation of PR or better, which was confirmed by a repeated measurement as required by the IMWG criteria.
Time Frame: From randomization to the date of initial documentation of PR or better (up to 5 years)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 98 | 100 | 16
Months | 0.8 [0.8 to 1.0] | 0.8 [0.8 to 0.8] | 0.8 [0.7 to 1.4]

13. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration from the date of randomization to the date of first documented evidence of progressive disease or death, whichever comes first. PD is defined as an increase of 25 % from the lowest response value in one of the following: serum and urine M-component (absolute increase must be >= 0.5 g/dL and >=200 mg/24 hours respectively); Only in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels (absolute increase must be > 10 mg/dL); Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: From randomization to the date of first documented evidence of progressive disease or death (up to 5 years)
Population: ITT analysis set which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 103 | 104 | 16
Months | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [57.6 to NA] — Here NA signifies that Median and upper limit of 95% CI was not estimable due to insufficient number of events.

14. Secondary Outcome: Overall Survival (OS)
Description: OS is measured from the date of randomization to the date of the participant's death.
Time Frame: From randomization to the date of initial documentation of participant's death (up to 5 years)
Population: ITT analysis set which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 103 | 104 | 16
Months | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events.

15. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the duration from the date of randomization to the date of first documented evidence of progressive disease according to the IMWG criteria.
Time Frame: From randomization to the date of first documented evidence of progressive disease (up to 5 years)
Population: ITT analysis set which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 103 | 104 | 16
Months | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [57.59 to NA] — Here NA signifies that Median and upper limit of 95% CI was not estimable due to insufficient number of events.

16. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the duration from the date of initial documentation of a response (PR or better) according to the IMWG criteria to the date of first documented evidence of progressive disease according to the IMWG criteria. PD is defined as an increase of 25 % from the lowest response value in one of the following: serum and urine M-component (absolute increase must be >= 0.5 g/dL and >=200 mg/24 hours respectively); Only in participants without measurable serum and urine M-protein levels the difference between involved and uninvolved FLC levels (absolute increase must be > 10 mg/dL); Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time Frame: From the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive (up to 5 years)
Population: Population analyzed included response evaluable analysis set who achieved response PR or better.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
Number analyzed (Participants) | 90 | 99 | 16
Months | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here NA signifies that Median and 95% CI was not estimable due to insufficient number of events. | NA [56.8 to NA] — Here NA signifies that Median and upper limit of 95% CI was not estimable due to insufficient number of events.

ADVERSE EVENTS:
Time Frame: Other adverse events and serious adverse events: up to 30 days after the last dose of study treatment (up to 3 years); All-cause mortality: up to end of study (up to 5 years)
Description: 4 participants in D-RVd and 2 in RVd group were randomized but did not receive any treatment. 1 participant in D-RVd group received RVd and was counted in D-RVd group for ITT and RVd group for safety analysis. So, safety analysis set (SAS) included 99 participants in D-RVd and 102 in RVd group. All-cause mortality was assessed in ITT set (included all randomized participants). SAEs and other AEs were assessed on SAS which included all participants who received at least 1 dose of study drugs.
Arm/Group | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) | Randomized: Daratumumab+RVd (D-RVd) | Safety Run-in: D-RVd
All-Cause Mortality (participants affected / at risk) | 7/103 | 7/104 | 1/16
Serious Adverse Events (participants affected / at risk) | 53/102 | 46/99 | 12/16
Other Adverse Events (participants affected / at risk) | 102/102 | 99/99 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) (N=102) | Randomized: Daratumumab+RVd (D-RVd) (N=99) | Safety Run-in: D-RVd (N=16)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0
Atrial Tachycardia (Cardiac disorders) | 1 | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0
Sickle Cell Anaemia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Infarction (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
Chest Pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 10 | 11 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 1 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Serum Sickness-Like Reaction (Immune system disorders) | 1 | 0 | 0
Acute Sinusitis (Infections and infestations) | 1 | 1 | 0
Adenovirus Infection (Infections and infestations) | 1 | 0 | 0
Aspergillus Infection (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Corona Virus Infection (Infections and infestations) | 0 | 1 | 0
Escherichia Infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Escherichia Coli (Infections and infestations) | 0 | 1 | 0
Gastroenteritis Salmonella (Infections and infestations) | 0 | 1 | 0
H1n1 Influenza (Infections and infestations) | 1 | 0 | 0
Herpes Zoster Disseminated (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 5 | 1 | 0
Parainfluenzae Virus Infection (Infections and infestations) | 1 | 0 | 0
Periorbital Abscess (Infections and infestations) | 0 | 1 | 0
Pneumococcal Bacteraemia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 14 | 15 | 5
Pneumonia Bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia Legionella (Infections and infestations) | 0 | 1 | 0
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 | 1 | 0
Rhinovirus Infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0
Septic Shock (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 1
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0
Clostridium Test Positive (Investigations) | 1 | 0 | 0
Human Rhinovirus Test Positive (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0
Neuralgia (Nervous system disorders) | 2 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 1 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0
Confusional State (Psychiatric disorders) | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 4 | 4 | 0
Bladder Perforation (Renal and urinary disorders) | 0 | 0 | 1
Glomerulonephritis Membranoproliferative (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Drug Reaction with Eosinophilia and Systemic Symptoms (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypersensitivity Vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized: Lenalidomide+Bortezomib+Dexamethasone (RVd) (N=102) | Randomized: Daratumumab+RVd (D-RVd) (N=99) | Safety Run-in: D-RVd (N=16)
Anaemia (Blood and lymphatic system disorders) | 33 | 37 | 7
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 30 | 39 | 10
Lymphopenia (Blood and lymphatic system disorders) | 29 | 31 | 13
Monocytosis (Blood and lymphatic system disorders) | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 41 | 63 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 36 | 44 | 8
Atrial Fibrillation (Cardiac disorders) | 3 | 2 | 0
Bradycardia (Cardiac disorders) | 2 | 3 | 1
Palpitations (Cardiac disorders) | 2 | 5 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 2 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 2 | 2
Tachycardia (Cardiac disorders) | 3 | 3 | 3
Ear Congestion (Ear and labyrinth disorders) | 1 | 2 | 0
Ear Discomfort (Ear and labyrinth disorders) | 0 | 3 | 0
Ear Pain (Ear and labyrinth disorders) | 2 | 3 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 3 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 9 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 1
Adrenal Insufficiency (Endocrine disorders) | 0 | 2 | 1
Hypothyroidism (Endocrine disorders) | 2 | 0 | 1
Cataract (Eye disorders) | 2 | 3 | 2
Dry Eye (Eye disorders) | 2 | 4 | 0
Eye Irritation (Eye disorders) | 3 | 1 | 0
Eye Swelling (Eye disorders) | 0 | 2 | 0
Lacrimation Increased (Eye disorders) | 2 | 4 | 1
Vision Blurred (Eye disorders) | 15 | 19 | 1
Visual Impairment (Eye disorders) | 1 | 2 | 0
Vitreous Floaters (Eye disorders) | 1 | 3 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 5 | 0
Abdominal Distension (Gastrointestinal disorders) | 4 | 8 | 3
Abdominal Pain (Gastrointestinal disorders) | 10 | 24 | 6
Abdominal Pain Lower (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 6 | 1
Constipation (Gastrointestinal disorders) | 42 | 51 | 6
Dental Caries (Gastrointestinal disorders) | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 56 | 65 | 10
Dry Mouth (Gastrointestinal disorders) | 6 | 7 | 1
Dyspepsia (Gastrointestinal disorders) | 10 | 15 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 3 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 11 | 1
Gingival Pain (Gastrointestinal disorders) | 0 | 2 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 2 | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 4 | 3 | 1
Nausea (Gastrointestinal disorders) | 51 | 51 | 6
Oral Dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 1
Oral Pain (Gastrointestinal disorders) | 1 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 5 | 3
Toothache (Gastrointestinal disorders) | 1 | 10 | 0
Vomiting (Gastrointestinal disorders) | 29 | 32 | 5
Asthenia (General disorders) | 9 | 3 | 1
Catheter Site Pain (General disorders) | 0 | 2 | 0
Chest Discomfort (General disorders) | 3 | 9 | 0
Chills (General disorders) | 9 | 26 | 4
Face Oedema (General disorders) | 1 | 4 | 2
Fatigue (General disorders) | 63 | 71 | 10
Gait Disturbance (General disorders) | 4 | 3 | 0
Influenza Like Illness (General disorders) | 8 | 18 | 0
Injection Site Erythema (General disorders) | 2 | 4 | 0
Injection Site Pruritus (General disorders) | 1 | 0 | 1
Injection Site Rash (General disorders) | 4 | 4 | 1
Injection Site Reaction (General disorders) | 3 | 4 | 0
Localised Oedema (General disorders) | 2 | 5 | 0
Malaise (General disorders) | 2 | 7 | 2
Non-Cardiac Chest Pain (General disorders) | 6 | 8 | 2
Oedema (General disorders) | 7 | 5 | 1
Oedema Peripheral (General disorders) | 37 | 36 | 6
Pain (General disorders) | 7 | 11 | 1
Peripheral Swelling (General disorders) | 3 | 10 | 1
Pyrexia (General disorders) | 27 | 43 | 7
Swelling (General disorders) | 0 | 1 | 1
Swelling Face (General disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 3 | 2
Hypersensitivity (Immune system disorders) | 1 | 2 | 1
Hypogammaglobulinaemia (Immune system disorders) | 0 | 3 | 3
Seasonal Allergy (Immune system disorders) | 2 | 5 | 0
Acute Sinusitis (Infections and infestations) | 0 | 3 | 0
Adenovirus Infection (Infections and infestations) | 0 | 2 | 0
Anal Tinea (Infections and infestations) | 0 | 0 | 1
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 1
Bacterial Infection (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 4 | 7 | 4
Candida Infection (Infections and infestations) | 2 | 2 | 0
Cellulitis (Infections and infestations) | 4 | 7 | 2
Conjunctivitis (Infections and infestations) | 3 | 6 | 1
Conjunctivitis Bacterial (Infections and infestations) | 0 | 0 | 1
Corona Virus Infection (Infections and infestations) | 1 | 3 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 1
Ear Infection (Infections and infestations) | 0 | 2 | 2
Eye Infection (Infections and infestations) | 1 | 2 | 1
Folliculitis (Infections and infestations) | 0 | 2 | 0
Furuncle (Infections and infestations) | 1 | 2 | 0
Gastroenteritis Viral (Infections and infestations) | 3 | 2 | 2
Gastrointestinal Infection (Infections and infestations) | 0 | 2 | 0
Gastrointestinal Viral Infection (Infections and infestations) | 0 | 2 | 0
Gingivitis (Infections and infestations) | 3 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 4 | 0
Hordeolum (Infections and infestations) | 3 | 4 | 0
Influenza (Infections and infestations) | 7 | 14 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 2
Metapneumovirus Infection (Infections and infestations) | 1 | 0 | 1
Nail Infection (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 4 | 12 | 2
Oral Candidiasis (Infections and infestations) | 2 | 3 | 0
Oral Herpes (Infections and infestations) | 0 | 2 | 0
Otitis Media (Infections and infestations) | 0 | 4 | 0
Parainfluenzae Virus Infection (Infections and infestations) | 2 | 5 | 1
Paronychia (Infections and infestations) | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 4 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 7 | 14 | 3
Pneumonia Influenzal (Infections and infestations) | 0 | 0 | 1
Rash Pustular (Infections and infestations) | 3 | 5 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 3 | 3 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 0
Rhinitis (Infections and infestations) | 1 | 2 | 0
Rhinovirus Infection (Infections and infestations) | 2 | 6 | 0
Sinusitis (Infections and infestations) | 8 | 13 | 3
Skin Infection (Infections and infestations) | 1 | 2 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 3 | 0
Tooth Infection (Infections and infestations) | 2 | 5 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 51 | 67 | 11
Urinary Tract Infection (Infections and infestations) | 5 | 11 | 2
Vaginal Infection (Infections and infestations) | 1 | 2 | 0
Viral Infection (Infections and infestations) | 0 | 1 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 5 | 7 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 2 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 7 | 12 | 1
Fall (Injury, poisoning and procedural complications) | 13 | 9 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 2 | 0
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 4 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 5 | 0
Vascular Access Site Swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1
Adjusted Calcium (Investigations) | 1 | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 18 | 18 | 1
Aspartate Aminotransferase Increased (Investigations) | 18 | 13 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 11 | 13 | 1
Blood Creatinine Increased (Investigations) | 7 | 8 | 0
Coronavirus Test Positive (Investigations) | 1 | 3 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 2
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 2 | 0
Haematocrit Decreased (Investigations) | 0 | 2 | 0
Human Rhinovirus Test Positive (Investigations) | 0 | 2 | 0
Protein Total Decreased (Investigations) | 1 | 5 | 0
Weight Decreased (Investigations) | 4 | 10 | 0
Weight Increased (Investigations) | 3 | 6 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 11 | 24 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 6 | 0
Gout (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 22 | 12 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 6 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 7 | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 | 11 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 17 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 27 | 28 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 | 9 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 15 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 17 | 15 | 5
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 | 3 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 38 | 39 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 35 | 41 | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 | 16 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 20 | 30 | 3
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 13 | 11 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 14 | 16 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 11 | 13 | 3
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 27 | 4
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 10 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 22 | 22 | 6
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2
Melanocytic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Amnesia (Nervous system disorders) | 3 | 4 | 0
Cerebral Congestion (Nervous system disorders) | 1 | 2 | 0
Cognitive Disorder (Nervous system disorders) | 1 | 3 | 0
Disturbance in Attention (Nervous system disorders) | 1 | 3 | 0
Dizziness (Nervous system disorders) | 25 | 23 | 2
Dizziness Postural (Nervous system disorders) | 1 | 3 | 0
Dysgeusia (Nervous system disorders) | 19 | 23 | 1
Headache (Nervous system disorders) | 24 | 33 | 3
Hyperaesthesia (Nervous system disorders) | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 6 | 5 | 0
Memory Impairment (Nervous system disorders) | 8 | 2 | 2
Migraine (Nervous system disorders) | 3 | 1 | 0
Neuralgia (Nervous system disorders) | 9 | 11 | 1
Neuropathy Peripheral (Nervous system disorders) | 43 | 25 | 2
Paraesthesia (Nervous system disorders) | 10 | 23 | 4
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 39 | 39 | 6
Presyncope (Nervous system disorders) | 3 | 2 | 0
Restless Legs Syndrome (Nervous system disorders) | 0 | 2 | 0
Sciatica (Nervous system disorders) | 3 | 0 | 0
Sinus Headache (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 4 | 5 | 1
Taste Disorder (Nervous system disorders) | 3 | 1 | 1
Tremor (Nervous system disorders) | 8 | 11 | 2
Agitation (Psychiatric disorders) | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 14 | 18 | 3
Confusional State (Psychiatric disorders) | 1 | 2 | 1
Depression (Psychiatric disorders) | 5 | 8 | 1
Insomnia (Psychiatric disorders) | 31 | 45 | 6
Irritability (Psychiatric disorders) | 1 | 2 | 0
Libido Decreased (Psychiatric disorders) | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 2 | 2 | 0
Sleep Disorder (Psychiatric disorders) | 3 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 5 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 2 | 0
Dysuria (Renal and urinary disorders) | 5 | 5 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 5 | 0
Polyuria (Renal and urinary disorders) | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 1
Renal Impairment (Renal and urinary disorders) | 4 | 2 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 2 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 3 | 4 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 3 | 0
Vaginal Fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 2 | 0
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 53 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 24 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 14 | 22 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 13 | 17 | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 1
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 5 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 10 | 13 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 5 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 7 | 4 | 3
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 4 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 18 | 1
Rash (Skin and subcutaneous tissue disorders) | 26 | 25 | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 25 | 24 | 3
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin Mass (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 5 | 0
Deep Vein Thrombosis (Vascular disorders) | 6 | 1 | 0
Embolism (Vascular disorders) | 3 | 2 | 0
Flushing (Vascular disorders) | 2 | 10 | 2
Hot Flush (Vascular disorders) | 5 | 8 | 0
Hypertension (Vascular disorders) | 15 | 12 | 6
Hypotension (Vascular disorders) | 13 | 9 | 1
Lymphoedema (Vascular disorders) | 0 | 1 | 1
Orthostatic Hypertension (Vascular disorders) | 0 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 3 | 5 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Initial protocol did not require minimal residual disease (MRD) testing in all participants, impacting the interpretation of MRD negativity rates in intent-to-treat (ITT) group, which strongly favored daratumumab treatment. Sensitivity analysis, including MRD negativity rate in participants with a complete response (CR) or better and with an informative baseline clone and follow-up MRD testing, were performed and confirmed a strong benefit for daratumumab treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT02874742/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/42/NCT02874742/SAP_001.pdf